CLINICAL TRIAL: NCT00833053
Title: A Study of Dose Optimization of Infliximab in the Treatment of Moderate to Severe Plaque Psoriasis
Brief Title: Dose Optimization of Infliximab in Moderate to Severe Plaque Psoriasis (Study P05315)
Acronym: DOSE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: In Amendment 1 of P05319 [NCT 00779675], the option to enroll into this study, was discontinued due to low numbers of participants with suboptimal response.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05315; EUDRACT: 2008-000454-12
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Results first posted 2012-07-26 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Infliximab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IFX q 6 weeks (Experimental)
  Interventions: Drug: Infliximab
- IFX + MTX (Experimental)
  Interventions: Drug: Infliximab and methotrexate

INTERVENTIONS:
Drug: Infliximab — Infliximab 5 mg/kg body weight intravenous infusion given every 6 weeks
  Other Names: Remicade; SCH 215596
  Arms: IFX q 6 weeks
Drug: Infliximab and methotrexate — Infliximab 5 mg/kg body weight intravenous infusion (given every 8 weeks) plus methotrexate 7.5 mg orally (once weekly)
  Other Names: Remicade; SCH 215596
  Arms: IFX + MTX

SUMMARY:
Participants from an ongoing observational study (P05319) who have a limited (adequate but less than optimal) response to infliximab will be randomized to either increase the frequency of infliximab infusions from every 8 weeks to every 6 weeks, or to add weekly methotrexate to their current treatment plan. While receiving infliximab study treatment(s), patients in this study will attend regularly scheduled office visits for various clinical tests for safety and effectiveness evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosis of moderate to severe plaque-type psoriasis and have had participated in Study P05319.
* Subjects must have demonstrated an adequate but suboptimal response to infliximab in Study P05319
* Subjects must be at least 18 years old
* Subjects must be candidates for phototherapy or systemic treatment for psoriasis.
* Subjects must not be pregnant and must meet contraceptive requirements
* Subjects must meet tuberculosis screening criteria
* Subjects must meet laboratory and medical history screening requirements

Exclusion Criteria:

* Subjects for whom infliximab or methotrexate is contraindicated or not recommended.
* Subjects already using certain investigational, biological, or immunosuppressive drugs
* Subjects with certain comorbid conditions
* Subjects who currently have or have a history of certain infections
* Subjects who have recently received live virus or bacterial vaccinations
* Subjects who are in a situation or have any condition that, in the opinion of the investigator, may interfere with optimal participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multicenter: 48 centers in Australia, Belgium, Colombia, Canada, Denmark, France, Germany, Greece, Hungary, Italy, and Russia.
Pre-assignment Details: Of the 39 participants that were randomized to the study, 3 (2 Infliximab [IFX] q 6 weeks; and 1 IFX + Methotrexate [MTX]) participants did not meet protocol eligibility criteria and were excluded from the efficacy analysis.
Groups:
- IFX q 6 Weeks: Infliximab 5 mg/kg administered every 6 weeks.
- IFX q 8 Weeks + MTX: Infliximab 5mg/kg administered every 8 weeks in combination with methotrexate 7.5 mg orally once weekly.
Period: Overall Study
Arm/Group | IFX q 6 Weeks | IFX q 8 Weeks + MTX
Started | 19 | 20
Completed | 10 | 17
Not Completed | 9 | 3
Not completed — Adverse Event | 4 | 0
Not completed — Treatment Failure | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IFX q 6 Weeks | IFX q 8 Weeks + MTX | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (15.38) | 48.2 (17.03) | 46.8 (16.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With A Psoriasis Area and Sensitivity Index (PASI)-75 Response at Week 28
Description: The Psoriasis Area and Sensitivity Index (PASI) is a measure of the average redness, thickness, and scaliness of psoriasis lesions. Each lesion is graded on a 0-4 scale, weighted by the area of involvement, with increasing scores indicating increasing severity. The PASI-75 response indicates the number of participants achieving a 75% reduction in PASI score compared to baseline.
Time Frame: Baseline, Week 28
Measure: Number; unit: Participants
Arm/Group | IFX q 6 Weeks | IFX q 8 Weeks + MTX
Number analyzed (Participants) | 17 | 19
Participants | 9 | 11

2. Secondary Outcome: Number of Participants With A PASI-50 Response at Week 28
Description: The PASI score is a measure of the average redness, thickness, and scaliness of psoriasis lesions. Each lesion is graded on a 0-4 scale, weighted by the area of involvement, with increasing scores indicating increasing severity.The PASI-50 response indicates the number of participants achieving a 50% reduction compared to baseline in PASI score.
Time Frame: Baseline, Week 28
Population: The study was terminated early with only 15% subjects of the original planned size. Accordingly, secondary efficacy analyses were cancelled due to such a small subject population.
Arm/Group | IFX q 6 Weeks | IFX q 8 Weeks + MTX
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With A PASI-90 Response at Week 28
Description: The PASI score is a measure of the average redness, thickness, and scaliness of psoriasis lesions. Each lesion is graded on a 0-4 scale, weighted by the area of involvement, with increasing scores indicating increasing severity. The PASI-90 response indicates the number of participants achieving a 90% reduction compared to baseline in PASI score.
Time Frame: Baseline, Week 28
Population: as for outcome 2
Arm/Group | IFX q 6 Weeks | IFX q 8 Weeks + MTX
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants With A PASI-100 Response at Week 28
Description: The PASI score is a measure of the average redness, thickness, and scaliness of psoriasis lesions. Each lesion is graded on a 0-4 scale, weighted by the area of involvement, with increasing scores indicating increasing severity. The PASI-100 response indicates the number of participants achieving a 100% reduction compared to baseline in PASI score.
Time Frame: Baseline, Week 28
Population: as for outcome 2
Arm/Group | IFX q 6 Weeks | IFX q 8 Weeks + MTX
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Mean Participant Raw PASI Scores at Week 28
Description: The PASI score is a measure of the average redness, thickness, and scaliness of psoriasis lesions. Each lesion is graded on a 0-4 scale, weighted by the area of involvement, with increasing scores indicating increasing severity.
Time Frame: Baseline, Week 28
Population: as for outcome 2
Arm/Group | IFX q 6 Weeks | IFX q 8 Weeks + MTX
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Dermatology Life Quality Index (DLQI) at Week 28
Description: The DLQI is a 10-item questionnaire. Scores range from 0-10 with 0 indicating high quality of life and 10 indicating poor quality of life.
Time Frame: Week 28
Population: as for outcome 2
Arm/Group | IFX q 6 Weeks | IFX q 8 Weeks + MTX
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Euro-Qol 5 Dimension (EQ-5D) Change From Baseline at Week 28
Description: The EQ-5D is a descriptive system comprised of the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Participants are asked to indicate his/her health state by selecting the most appropriate statement in each of the 5 dimensions. This selection results in a 1-digit number expressing the level selected for that dimension. The digits for 5 dimensions can be combined in a 5-digit number describing the participant's health state. The numerals 1-5 have no arithmetic properties and should not be used as a cardinal score.
Time Frame: Baseline, Week 28
Population: as for outcome 2
Arm/Group | IFX q 6 Weeks | IFX q 8 Weeks + MTX
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Safety analyses were performed on all randomized subjects who took at least one dose of study medication.
Arm/Group | IFX q 6 Weeks | IFX q 8 Weeks + MTX
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/19
Other Adverse Events (participants affected / at risk) | 8/18 | 6/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IFX q 6 Weeks (N=18) | IFX q 8 Weeks + MTX (N=19)
Psoriasis Aggravated (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IFX q 6 Weeks (N=18) | IFX q 8 Weeks + MTX (N=19)
Vertigo (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Duodenal Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest Discomfort (General disorders) | 1 (1) | 0 (0)
Infusion Related Reaction (General disorders) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Oral Herpes (Infections and infestations) | 1 (2) | 0 (0)
Rash Pustular (Infections and infestations) | 0 (0) | 1 (1)
Renal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (4)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Arthropod Sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood Pressure Increased (Investigations) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscle Spasm (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Hypotonia (Nervous system disorders) | 1 (1) | 0 (0)
Vaginal Inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus Generalized (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less